CLINICAL TRIAL: NCT01734590
Title: The Effect of Different Flour Compositions in a Carbohydrate-based Food on Rate of Exogenous Glucose Appearance in Blood.
Brief Title: Effect of Different Flour Compositions in a Carbohydrate-based Food on Rate of Exogenous Glucose Appearance in Blood
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Unilever R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: FDS-NAA-0758
Record Dates: First submitted 2012-11-21; First posted 2012-11-27 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Healthy
Keywords: Flour,; carbohydrate,; digestibility; subjects

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- Carbohydrate based food mix 1 (Experimental): Slowly digestible carbohydrate
  Interventions: Dietary Supplement: Carbohydrate based food mix 2; Dietary Supplement: Control carbohydrate based food
- Carbohydrate based food mix 2 (Experimental): Slowly digestible carbohydrate
  Interventions: Dietary Supplement: Carbohydrate based food mix 1; Dietary Supplement: Control carbohydrate based food
- Control carbohydrate based food (Active Comparator): Rapidly digestible carbohydrate
  Interventions: Dietary Supplement: Carbohydrate based food mix 1; Dietary Supplement: Carbohydrate based food mix 2

INTERVENTIONS:
Dietary Supplement: Carbohydrate based food mix 1 — Carbohydrate based food
  Other Names: Slowly digestible carbohydrate
  Arms: Carbohydrate based food mix 2; Control carbohydrate based food
Dietary Supplement: Carbohydrate based food mix 2 — Carbohydrate based food
  Other Names: Slowly digestible carbohydrate
  Arms: Carbohydrate based food mix 1; Control carbohydrate based food
Dietary Supplement: Control carbohydrate based food — Carbohydrate based food
  Other Names: Rapidly digestible carbohydrate
  Arms: Carbohydrate based food mix 1; Carbohydrate based food mix 2

SUMMARY:
Exploratory study with double-blind, randomized, placebo-controlled, full cross-over design.

The main objective is to identify one or two flour compositions in a carbohydrate-based food that produce a significant difference (alpha =0.2) in the time to reach 50% of cumulative absorption of exogenous glucose compared to the control.

DETAILED DESCRIPTION:
Twelve volunteers will participate in the study; each person will be studied on three different occasions at least one week apart, consuming the three different test products in a randomized order. Test products are carbohydrate-based food made from different flour mixes differing in their expected rate of intestinal starch digestion. The products are labeled with 13C starch.

ELIGIBILITY:
* healthy males
* Age at start of the study ≥18 and ≤ 50 years
* Not smoking
* Body mass index (BMI) ≥ 20 and ≤ 28 kg/m2
* Fasting blood glucose value of volunteer is ≥ 3.4 and ≤ 6.1 mmol/litre (i.e. 62-110 mg/dl) at screening

Ages: 18 Years to 50 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 12 (Actual)
Dates: Start 2012-11; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Rate of appearance of exogenous glucose (RaE) based on the dual isotope technique. | Measured during 360 min for 3 periods

SECONDARY OUTCOMES:
Total blood glucose and insulin | Measured during 360 min for 3 periods

CONTACTS AND LOCATIONS:
Overall Officials: Khalid Abd-Elaziz, Principal Investigator — QPS Netherlands BV
Locations (1):
- QPS, Groningen, Hanzeplein 1, Netherlands